CLINICAL TRIAL: NCT02565511
Title: A Randomized, Double-blind, Placebo-controlled, Two-cohort, Parallel Group Study to Evaluate the Efficacy of CAD106 and CNP520 in Participants at Risk for the Onset of Clinical Symptoms of Alzheimer's Disease.
Brief Title: A Study of CAD106 and CNP520 Versus Placebo in Participants at Risk for the Onset of Clinical Symptoms of Alzheimer's Disease
Acronym: GS1
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Banner Alzheimer's Institute (Other); National Institute on Aging (NIA) (NIH); Amgen (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAPI015A2201J; 2015-002715-15 (EudraCT Number); 1UF1AG046150-01 (NIH)
Record Dates: First submitted 2015-09-28; First posted 2015-10-01 (Estimated); Results first posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Alzheimers Disease
Keywords: Randomization; Placebo controlled; Parallel-group; APOE4 Homozygotes; Preclinical Alzheimers Disease (AD); Aβ lowering; CNP520; CAD106; elderly; Brain Amyloid; BACE-1 inhibitor; Prevention; Unimpaired cognition
MeSH Terms: conditions — Alzheimer Disease | interventions — Umibecestat; aluminum sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort I (CAD106) (Experimental): CAD106 (450 µg) + Alum (450 µg) intra-muscular injection at Weeks 1, 7, 13 and every 13 weeks thereafter
  Interventions: Biological: CAD106 Immunotherapy; Other: Alum
- Cohort I (CAD106 Placebo) (Placebo Comparator): Placebo to CAD106 + Alum (450 µg) intra-muscular injection at Weeks 1, 7, 13 and every 13 weeks thereafter
  Interventions: Other: Placebo to CAD106; Other: Alum
- Cohort II (CNP520) (Experimental): CNP520 (50 mg) capsules taken orally once daily
  Interventions: Drug: CNP520
- Cohort II (CNP520 Placebo) (Placebo Comparator): Matching Placebo to CNP520 capsules taken orally once daily
  Interventions: Other: Placebo to CNP520

INTERVENTIONS:
Biological: CAD106 Immunotherapy — Participants will be given i.m. injections at Weeks 1, 7, 13 and quarterly i.m. injections (every 13 weeks) thereafter, until the last injection 3 month prior to completion of the Treatment Epoch.
  Arms: Cohort I (CAD106)
Other: Placebo to CAD106 — Participants will be given i.m. injections at Weeks 1, 7, 13 and quarterly i.m. injections (every 13 weeks) thereafter, until the last injection 3 month prior to completion of the Treatment Epoch.
  Arms: Cohort I (CAD106 Placebo)
Drug: CNP520 — CNP520 50 mg capsule p.o. for the duration of the Treatment Epoch.
  Arms: Cohort II (CNP520)
Other: Placebo to CNP520 — Placebo to CNP520 p.o. for the duration of the Treatment Epoch
  Arms: Cohort II (CNP520 Placebo)
Other: Alum — Alum was mixed with reconstituted CAD106 as adjuvant therapy to maximize the effectiveness of CAD106
  Arms: Cohort I (CAD106 Placebo); Cohort I (CAD106)

SUMMARY:
The purpose of this study was to test whether two investigational drugs called CAD106 and CNP520, administered separately, could slow down the onset and progression of clinical symptoms associated with Alzheimer's disease (AD) in participants at the risk to develop clinical symptoms based on their age and genotype.

DETAILED DESCRIPTION:
The study (also known as the Generation Study 1, GS1) was conducted as part of the Alzheimer's Prevention Initiative (API) program.

This trial was a randomized, double-blind, placebo-controlled, parallel group, adaptive design with variable treatment duration planned in cognitively unimpaired APOE4 homozygotes (HMs) aged 60 to 75 years. Participants were enrolled into Cohort I (CAD106) or Cohort II (CNP520).

The planned treatment period of 5 to 8 years was not achieved due to early study termination.

The study was terminated due to unexpected changes in cognitive function, brain volume loss, and body weight loss. Cohort II (CNP520) treatment was stopped and evaluated through an off-treatment follow-up period. After the decision to terminate Cohort II of the study (CNP520), treatment with CAD106 (Cohort I) was also terminated.

ELIGIBILITY:
Key Inclusion Criteria:

* Consented to receive disclosure of their risk estimates to develop clinical symptoms of AD based on their APOE genotype.
* Male or female, age 60 to 75 years inclusive. Females were to be post-menopausal.
* Mini-Mental State Examination (MMSE) total score ≥ 24 and cognitively unimpaired as evaluated by memory tests
* Homozygous APOE4 genotype.
* Participant willing to have a study partner.

Key Exclusion Criteria:

* Any disability that prevented the participant from completing all study requirements.
* Current medical or neurological condition that could have impacted cognition or performance on cognitive assessments.
* Advanced, severe progressive or unstable disease that may have interfered with the safety, tolerability and study assessments, or put the participant at special risk.
* History of malignancy of any organ system, treated or untreated, within 60 months prior to screening.
* History of hypersensitivity to any of the investigational drugs or their excipients / adjuvant or to drugs of similar chemical classes.
* Indication or on current treatment with ChEIs and/or another AD treatment (e.g. memantine).
* Contraindication or intolerance to MRI or PET investigations (with fluorinated radio ligands).
* Brain MRI results showing findings unrelated to AD that, in the opinion of the Investigator could have been a leading cause to future cognitive decline, pose a risk to the participant, or prevent a satisfactory MRI assessment for safety monitoring.
* Suicidal Ideation in the past six months or Suicidal Behavior in the past two years, prior to screening.
* A positive drug screen at Screening, if, in the Investigator's opinion, this was due to drug abuse.
* Significantly abnormal laboratory results at Screening, or infection not as a result of a temporary condition.
* Current clinically significant ECG findings. For Cohort - I only: Participants with previous organ transplantation or stem cell transplantation, or indication for treatment with anti-coagulants.

For Cohort - II only: Participants with depigmenting or hypopigmenting conditions (e.g. albinism vitiligo) or active / history of chronic urticarial in the past year.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (121):
- United States (77):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Scottsdale, Arizona
  - Banner Sun City Research Institute, Sun City, Arizona
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Irvine Center for Clinical Research, Irvine, California
  - University of Southern California Keck School of Medicine Alzheimer Disease Research Center, Los Angeles, California
  - Novartis Investigative Site, Palo Alto, California
  - Novartis Investigative Site, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - Novartis Investigative Site, Sebastopol, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - Novartis Investigative Site, Temecula, California
  - Novartis Investigative Site, Basalt, Colorado
  - Yale University Alzheimer's Disease Research Unit, New Haven, Connecticut
  - New England Institute for Clinical Research, Stamford, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - JEM Research Institute, Atlantis, Florida
  - Florida Atlantic University, Clinical Translational Research Unit, Boca Raton, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Meridien Research, Maitland, Florida
  - Merritt Island Medical Research, Merritt Island, Florida
  - University of Miami, Miami, Florida
  - Mount Sinai Medical Center - The Wien Center, Miami Beach, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Compass Research, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - USF Health Byrd Alzheimer's Institute, Tampa, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Medical Research & Health Education Foundation, Inc., Columbus, Georgia
  - NeuroStudies, Decatur, Georgia
  - Advanced Clinical Research, Meridian, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Alzheimer's Disease Center, Fairway, Kansas
  - Via Christi Research, Wichita, Kansas
  - Sanders Brown Center on Aging, University of Kentucky, Lexington, Kentucky
  - Novartis Investigative Site, Bangor, Maine
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Kalamazoo, Michigan
  - Novartis Investigative Site, Saint Paul, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Memory Disorders Program, Department of Neurological Sciences, University of Nebraska Medical Center, Omaha, Nebraska
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Memory Enhancement Center, Eatontown, New Jersey
  - The Memory Center of Northeastern New York, Latham, New York
  - NYU Langone Medical Center, New York, New York
  - The Nathan S. Kline Institute, Orangeburg, New York
  - University of Rochester Medical Center, Rochester, New York
  - Alzheimer's Memory Center, Charlotte, North Carolina
  - Duke University Medical center, Durham, North Carolina
  - Triad Clinical Trials, LLC, Greensboro, North Carolina
  - University Hospitals Cleveland Medical Center / Case Western Reserve University, Beachwood, Ohio
  - Novartis Investigative Site, Centerville, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Memory Health Center at Summit Research Network, Portland, Oregon
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Abington Neurological Associates, Willow Grove, Pennsylvania
  - Butler Hospital Memory and Aging Program, Providence, Rhode Island
  - Roper St. Francis - CBRI, Charleston, South Carolina
  - Novartis Investigative Site, Knoxville, Tennessee
  - CNS Healthcare, Memphis, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Senior Adults Specialty Research, Austin, Texas
  - Kerwin Research Center & Memory Care, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas Health Science Center, Houston, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - The Memory Clinic, Bennington, Vermont
  - Universal Research Group, Tacoma, Washington
  - The Medical College of WI, Milwaukee, Wisconsin
- Australia (3):
  - Novartis Investigative Site, Darlinghurst, New South Wales
  - Novartis Investigative Site, Heidelberg Heights, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Belgium (2):
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Canada (10):
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - Novartis Investigative Site, Kentville, Nova Scota
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, London, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - The Centre for Memory and Aging, Toronto, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Gatineau, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
- Novartis Investigative Site, Turku, Finland
- Germany (12):
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Böblingen
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Wenzenbach
- Novartis Investigative Site, Amsterdam, Netherlands
- Spain (4):
  - Novartis Investigative Site, Terrassa, Barcelona
  - Novartis Investigative Site, Pozuelo de Alarcón, Madrid
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Donostia / San Sebastian
- Novartis Investigative Site, Basel, CH, Switzerland
- United Kingdom (10):
  - Novartis Investigative Site, Westbruy on Trym, Bristol
  - Novartis Investigative Site, Exeter, Devon
  - Novartis Investigative Site, Plymouth, Devon
  - Novartis Investigative Site, Guildford, Surrey
  - Novartis Investigative Site, Avon
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Dundee
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 713 participants were screened
Groups:
- Cohort I (CI) CAD106: CAD106 (450 µg) + Alum (450 µg) intra-muscular injection at Weeks 1, 7, 13 and every 13 weeks thereafter
- Cohort I (CI) CAD106 Placebo: Placebo to CAD106 + Alum (450 µg) intra-muscular injection at Weeks 1, 7, 13 and every 13 weeks thereafter
- Cohort II (CII) CNP520: CNP520 (50 mg) capsules taken once daily orally
- Cohort II (CII) CNP520 Placebo: Placebo to CNP520 capsules taken once daily orally
Period: Overall Study
Arm/Group | Cohort I (CI) CAD106 | Cohort I (CI) CAD106 Placebo | Cohort II (CII) CNP520 | Cohort II (CII) CNP520 Placebo
Started | 42 | 23 | 251 | 164
3 Patients Were Mis-randomized | 0 | 0 | 2 | 1
Completed | 0 | 0 | 0 | 0
Not Completed | 42 | 23 | 251 | 164
Not completed — Study terminated by Sponsor | 35 | 22 | 235 | 156
Not completed — Withdrawal by Subject | 3 | 0 | 12 | 5
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 4 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Protocol deviation | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Three participants were included in the Participant Flow in Cohort II but not included in Baseline Characteristics because they were mis-randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I (CI) CAD106 | Cohort I (CI) CAD106 Placebo | Cohort II (CII) CNP520 | Cohort II (CII) CNP520 Placebo | Total
Number analyzed (Participants) | 42 | 23 | 249 | 163 | 477
Age, Customized [Number; unit: participants]
  <=64 years | 20 | 9 | 77 | 52 | 158
  65-69 years | 18 | 7 | 116 | 65 | 206
  >70 years | 4 | 7 | 56 | 46 | 113
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 17 | 129 | 102 | 275
  Male | 15 | 6 | 120 | 61 | 202
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 41 | 22 | 241 | 162 | 466
  Black | 1 | 1 | 1 | 0 | 3
  Asian | 0 | 0 | 4 | 0 | 4
  Pacific Islander | 0 | 0 | 1 | 0 | 1
  Other | 0 | 0 | 1 | 0 | 1
  Unknown | 0 | 0 | 1 | 1 | 2
Cohort I API Preclinical Composite Cognitive Battery (APCC) [Mean (Standard Deviation); unit: Scores on a scale] — APCC (API Preclinical Compo site Cognitive Battery) is a composite score derived from RBANS (Repeatable Battery for Assessment of Neurological Status), MMSE (Mini-Mental State Examination) and the Raven's Progressive Matrices; scores are 0-100 and higher scores indicate better cognitive performance. Population: Numbers in row represent participants in either Cohort I or Cohort II
  Scores on a scale
    number analyzed (Participants) | 42 | 23 | 0 | 0 | 65
    (all) | 78.0 (5.53) | 79.0 (6.76) |  |  | 78.3 (5.96)
Cohort I Repeatable Battery for Assessment of Neurological Status (RBANS) [Mean (Standard Deviation); unit: Scores on a scale] — RBANS is a tool to detect/characterize neurocognitive dementia changes in 5 neurocognitive domains; scores are 40-160 and higher scores indicate better cognitive functioning. Population: Numbers in row represent participants in either Cohort I or Cohort II
  Scores on a scale
    number analyzed (Participants) | 42 | 23 | 0 | 0 | 65
    (all) | 104.4 (12.03) | 108.7 (12.83) |  |  | 106.0 (12.39)
Cohort I Clinical Dementia Rating Sum of Boxes (CDR-SOB) [Mean (Standard Deviation); unit: scores on a scale] — Clinical Dementia Rating Sum of Boxes (CDR-SOB) measures cognition and functioning in 6 domains; scores are : 0-18 and higher scores indicate greater disease severity Population: Numbers in row represent participants in either Cohort I or Cohort II
  scores on a scale
    number analyzed (Participants) | 42 | 23 | 0 | 0 | 65
    (all) | 0.10 (0.276) | 0.04 (0.209) |  |  | 0.08 (0.254)
Cohort II API Preclinical Composite Cognitive Battery (APCC) [Mean (Standard Deviation); unit: scores on a scale] — Assessment of Neurological Status), MMSE(Mini-Mental State Examination) and the Raven's Progressive Matrices; scores are 0-100 and higher scores indicate better cognitive APCC(API Preclinical Composite Cognitive Battery) is a composite score derived from RBANS(Repeatable Battery for performance Population: Numbers in row represent participants in either Cohort I or Cohort II
  scores on a scale
    number analyzed (Participants) | 0 | 0 | 249 | 163 | 412
    (all) |  |  | 29.0 (1.17) | 28.9 (1.33) | 29.0 (1.23)
Cohort II Repeatable Battery for Assessment of Neurological Status (RBANS) [Mean (Standard Deviation); unit: scores on a scale] — RBANS is a tool to detect/characterize neurocognitive dementia changes in 5 neurocognitive domains; scores are 40-160 and higher scores indicate better cognitive functioning Population: Numbers in row represent participants in either Cohort I or Cohort II
  scores on a scale
    number analyzed (Participants) | 0 | 0 | 249 | 163 | 412
    (all) |  |  | 102.6 (12.22) | 103.2 (12.03) | 102.9 (12.13)
Cohort II Clinical Dementia Rating Sum of Boxes (CDR-SOB) [Mean (Standard Deviation); unit: scores on a scale] — Clinical Dementia Rating Sum of Boxes (CDR-SOB) measures cognition and functioning in 6 domains; scores are : 0-18 and higher scores indicate greater disease severity Population: Numbers in row represent participants in either Cohort I or Cohort II
  scores on a scale
    number analyzed (Participants) | 0 | 0 | 249 | 163 | 412
    (all) |  |  | 0.16 (0.15) | 0.15 (0.417) | 0.16 (0.409)

OUTCOME MEASURES:

1. Primary Outcome: Time to Event (Diagnosis of Mild Cognitive Impairment or Dementia, Due to Alzheimer's Disease (AD))
Description: Event was defined as the first confirmed diagnosis of MCI due to Alzheimer's disease (AD) or dementia due to AD (whichever occurred first) after adjudication by the progression adjudication committee (PAC) as triggered either by an investigator diagnosis or an increase in the Clinical Dementia Rating (CDR) global score. An event had to be confirmed by the PAC at two consecutive visits. In case no confirmed event was observed for a participant, the observation was censored, and the censoring date was defined as the last date where the diagnostic classification was assessed. The Study was terminated and only confirmed events collected up to the data cut-off point were counted. Due to the early termination of the study only a small number of events were observed and time-to-event could not be analyzed. Kaplan-Meyer (KM) estimates were provided to estimate probability that a subject would have an event prior to the specified visit.
Time Frame: Baseline to end of exposure for a maximum of 1455 days for CI and 907 days for CII
Population: n=number of participants at risk to experience an event at the time-point
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort I (CI) CAD106 | Cohort I (CI) CAD106 Placebo | Cohort II (CII) CNP520 | Cohort II (CII) CNP520 Placebo
Number analyzed (Participants) | 41 | 22 | 193 | 126
proportion of participants
  Week 26 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00] | 0.98 [0.95 to 0.99] | 0.98 [0.94 to 0.99]
  Week 52: number analyzed (Participants) | 40 | 22 | 95 | 63
  Week 52 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00] | 0.93 [0.88 to 0.96] | 0.95 [0.90 to 0.98]
  Week 78: number analyzed (Participants) | 37 | 21 | 18 | 9
  Week 78 | 0.97 [0.83 to 1.00] | 1.00 [1.00 to 1.00] | 0.88 [0.79 to 0.93] | 0.85 [0.63 to 0.94]
  Week 104: number analyzed (Participants) | 22 | 15 | 5 | 2
  Week 104 | 0.97 [0.83 to 1.00] | 1.00 [1.00 to 1.00] | 0.88 [0.79 to 0.93] | 0.85 [0.63 to 0.94]

2. Primary Outcome: Change in the Alzheimer's Prevention Initiative Composite Cognitive (APCC) Test Score
Description: APCC is a composite score derived from the specific scores from the Repeatable Battery for the Assessment of Neurological Status (RBANS), Mini-Mental State Examination (MMSE) and the Raven's Progressive Matrices. The APCC score is a weighted score with ranges from from 0 to 100 where higher scores correspond to better cognitive performance.
Time Frame: CI = Baseline to Weeks 26, 52,78 104 and Baseline to last assessment; CII = Baseline to Weeks 26, 52, 78, 104 and Baseline to Last on-treatment and Baseline to Last off-treatment
Population: Only participants with a value at both Baseline and that visit are included. For CI: last post-baseline assessment collected during the study. For CII: Last on-treatment is the last assessment before or at last day on study drug + 31 days. Last off-treatment is the last assessment after last day on study drug + 31 days.
Measure: Mean (Standard Deviation); unit: Total scores
Arm/Group | Cohort I (CI) CAD106 | Cohort I (CI) CAD106 Placebo | Cohort II (CII) CNP520 | Cohort II (CII) CNP520 Placebo
Number analyzed (Participants) | 41 | 23 | 179 | 125
Total scores
  Week 26: number analyzed (Participants) | 41 | 23 | 154 | 105
  Week 26 | -1.1 (4.10) | -2.0 (3.90) | -3.3 (4.54) | -1.0 (4.65)
  Week 52: number analyzed (Participants) | 41 | 22 | 64 | 36
  Week 52 | 0.9 (4.24) | 1.4 (3.36) | 0.3 (4.27) | 2.2 (6.11)
  Week 78: number analyzed (Participants) | 27 | 18 | 7 | 8
  Week 78 | 0.2 (4.15) | -0.7 (5.48) | -4.1 (4.14) | 2.4 (4.23)
  Week 104: number analyzed (Participants) | 17 | 9 | 3 | 0
  Week 104 | -1.4 (4.67) | 0.3 (4.00) | -6.7 (3.95) |
  CI-Last post BL assessment: number analyzed (Participants) | 41 | 23 | 0 | 0
  CI-Last post BL assessment | 0.0 (4.62) | 0.1 (3.87) |  |
  CII - Last on treatment: number analyzed (Participants) | 0 | 0 | 179 | 125
  CII - Last on treatment |  |  | -1.7 (4.81) | 0.1 (4.58)
  CII-Last off treatment: number analyzed (Participants) | 0 | 0 | 166 | 90
  CII-Last off treatment |  |  | -0.1 (4.72) | 0.2 (4.56)

3. Secondary Outcome: Change in Clinical Dementia Rating Scale Sum of Boxes (CDR-SOB) Score
Description: The CDR was obtained through semi-structured interviews of participants and informants, and cognitive functioning was rated on a 5-point scale of functioning in six domains: memory, orientation, judgement and problem solving, community affairs, home and hobbies, and personal care. The CDR global score ranged from zero to three, while the CDR-SOB was the sum of the ratings from the six domains, ranging from 0 to 18 with a minimum increment of 0.5. Higher scores indicated greater disease severity.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cohort I (CI) CAD106 | Cohort I (CI) CAD106 Placebo | Cohort II (CII) CNP520 | Cohort II (CII) CNP520 Placebo
Number analyzed (Participants) | 41 | 23 | 174 | 122
Scores on a scale
  Week 26: number analyzed (Participants) | 41 | 23 | 153 | 105
  Week 26 | -0.04 (0.234) | 0.00 (0.000) | 0.04 (0.361) | 0.00 (0.336)
  Week 52: number analyzed (Participants) | 41 | 23 | 64 | 36
  Week 52 | -0.01 (0.237) | 0.02 (0.104) | -0.02 (0.281) | -0.08 (0.541)
  Week 78: number analyzed (Participants) | 27 | 18 | 7 | 7
  Week 78 | -0.04 (0.237) | 0.03 (0.118) | 0.14 (0.802) | -0.14 (0.244)
  Week 104: number analyzed (Participants) | 17 | 9 | 3 | 0
  Week 104 | 0.15 (0.460) | 0.06 (0.167) | -0.17 (0.764) |
  CI Last post baseline assessment: number analyzed (Participants) | 41 | 23 | 0 | 0
  CI Last post baseline assessment | 0.04 (0.343) | 0.00 (0.302) |  |
  CII Last on-treatment: number analyzed (Participants) | 0 | 0 | 174 | 122
  CII Last on-treatment |  |  | 0.06 (0.505) | 0.03 (0.410)
  CII Last off-treatment: number analyzed (Participants) | 0 | 0 | 156 | 90
  CII Last off-treatment |  |  | 0.05 (0.464) | -0.01 (0.519)

4. Secondary Outcome: Change in the Total Scores of the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS).
Description: Repeatable Battery for the Assessment of Neurological Status (RBANS) is a clinical tool designed to detect and characterize the earliest neurocognitive changes associated with dementia. The RBANS generates age-adjusted index scores for five neurocognitive domains: Immediate Memory, Visuospatial/Constructional, Language, Attention and Delayed Memory, which are used to calculate a Total Scale Index score. Index scores and total score range from 40 to 160 and a higher score indicates better cognitive functioning.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | Cohort I (CI) CAD106 | Cohort I (CI) CAD106 Placebo | Cohort II (CII) CNP520 | Cohort II (CII) CNP520 Placebo
Number analyzed (Participants) | 41 | 23 | 209 | 141
scores
  Total Week 26: number analyzed (Participants) | 41 | 23 | 154 | 105
  Total Week 26 | -5.1 (7.25) | -3.0 (7.51) | -4.1 (8.58) | -2.6 (7.83)
  Total Week 52: number analyzed (Participants) | 41 | 22 | 64 | 37
  Total Week 52 | -1.2 (7.82) | 4.5 (7.10) | -0.1 (7.91) | 1.4 (8.06)
  Total Week 78: number analyzed (Participants) | 27 | 18 | 7 | 8
  Total Week 78 | -2.1 (7.69) | -4.0 (7.82) | -12.1 (7.40) | -4.8 (5.99)
  Total Week 104: number analyzed (Participants) | 17 | 9 | 3 | 0
  Total Week 104 | -1.4 (6.74) | -3.0 (8.34) | -7.7 (15.57) |
  Total CI Last post baseline assessment: number analyzed (Participants) | 41 | 23 | 0 | 0
  Total CI Last post baseline assessment | -1.0 (9.27) | 0.4 (7.20) |  |
  Total CII Last on-treatment: number analyzed (Participants) | 0 | 0 | 209 | 141
  Total CII Last on-treatment |  |  | -2.7 (8.65) | -0.2 (9.22)
  Total CII Last off-treatment: number analyzed (Participants) | 0 | 0 | 169 | 93
  Total CII Last off-treatment |  |  | -1.5 (9.20) | -0.6 (8.83)

5. Secondary Outcome: Change in the Index Scores of the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS).
Description: as for outcome 4
Time Frame: CI = Baseline to Weeks 26, 52 and Baseline to last assessment; CII = Baseline to Weeks 26, 52 and Baseline to Last on-treatment and Baseline to Last off-treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | Cohort I (CI) CAD106 | Cohort I (CI) CAD106 Placebo | Cohort II (CII) CNP520 | Cohort II (CII) CNP520 Placebo
Number analyzed (Participants) | 41 | 23 | 209 | 141
scores
  Immediate memory - Week 26: number analyzed (Participants) | 41 | 23 | 154 | 105
  Immediate memory - Week 26 | -8.6 (10.68) | -3.8 (11.16) | -7.4 (13.11) | -3.7 (12.15)
  Immediate memory - Week 52: number analyzed (Participants) | 41 | 22 | 64 | 37
  Immediate memory - Week 52 | 1.3 (10.81) | 4.8 (8.68) | 0.6 (13.55) | 5.1 (11.73)
  CI Immediate memory - Last post baseline assessment: number analyzed (Participants) | 41 | 23 | 0 | 0
  CI Immediate memory - Last post baseline assessment | -1.1 (13.11) | 1.1 (14.52) |  |
  CII Immediate memory - Last on-treatment: number analyzed (Participants) | 0 | 0 | 209 | 141
  CII Immediate memory - Last on-treatment |  |  | -3.7 (14.43) | 0.6 (13.54)
  CII Immediate memory - Last off-treatment: number analyzed (Participants) | 0 | 0 | 169 | 93
  CII Immediate memory - Last off-treatment |  |  | -3.2 (13.76) | -2.0 (11.90)
  Visuospatial Week 26: number analyzed (Participants) | 41 | 23 | 154 | 105
  Visuospatial Week 26 | -6.5 (15.21) | 0.7 (12.39) | -3.5 (14.98) | -2.4 (13.00)
  Visuospatial Week 52: number analyzed (Participants) | 41 | 22 | 64 | 37
  Visuospatial Week 52 | -6.5 (14.59) | 3.0 (15.09) | -1.4 (14.29) | -4.8 (12.60)
  CI Visuospatial Last post baseline assessment: number analyzed (Participants) | 41 | 23 | 0 | 0
  CI Visuospatial Last post baseline assessment | -4.7 (13.91) | 1.9 (12.72) |  |
  CII Visuospatial Last on-treatment n=: number analyzed (Participants) | 0 | 0 | 209 | 141
  CII Visuospatial Last on-treatment n= |  |  | -3.5 (14.59) | -2.6 (14.92)
  CII Visuospatial Last off-treatment: number analyzed (Participants) | 0 | 0 | 169 | 93
  CII Visuospatial Last off-treatment |  |  | -1.2 (15.13) | -0.8 (15.18)
  Language Week 26: number analyzed (Participants) | 41 | 23 | 154 | 105
  Language Week 26 | -1.4 (12.91) | -2.8 (11.42) | -0.1 (12.05) | -1.5 (11.87)
  Language Week 52: number analyzed (Participants) | 41 | 22 | 64 | 37
  Language Week 52 | 2.6 (10.29) | 2.0 (11.51) | -0.3 (12.88) | 0.8 (9.72)
  CI Language Last post baseline assessment: number analyzed (Participants) | 41 | 23 | 0 | 0
  CI Language Last post baseline assessment | 1.9 (13.00) | -4.5 (12.86) |  |
  CII Language Last on-treatment: number analyzed (Participants) | 0 | 0 | 209 | 141
  CII Language Last on-treatment |  |  | -0.1 (12.07) | -0.1 (11.93)
  CII Language Last off-treatment: number analyzed (Participants) | 0 | 0 | 169 | 93
  CII Language Last off-treatment |  |  | -1.0 (13.19) | -1.8 (11.25)
  Attention Week 26: number analyzed (Participants) | 41 | 23 | 154 | 105
  Attention Week 26 | 1.8 (9.40) | -0.6 (14.19) | -0.7 (10.42) | -0.6 (11.67)
  Attention Week 52: number analyzed (Participants) | 41 | 22 | 64 | 37
  Attention Week 52 | 0.9 (10.80) | -0.5 (13.09) | -0.2 (10.02) | 2.7 (10.77)
  CI Attention Last post baseline assessment: number analyzed (Participants) | 41 | 23 | 0 | 0
  CI Attention Last post baseline assessment | 2.0 (12.91) | 2.0 (10.25) |  |
  CII Attention Last on-treatment: number analyzed (Participants) | 0 | 0 | 209 | 141
  CII Attention Last on-treatment |  |  | 0.1 (10.80) | 0.8 (11.20)
  CII-Attention Last off-treatment: number analyzed (Participants) | 0 | 0 | 169 | 93
  CII-Attention Last off-treatment |  |  | 1.0 (1.64) | 1.2 (11.07)
  Delayed memory - Week 26: number analyzed (Participants) | 41 | 23 | 154 | 105
  Delayed memory - Week 26 | -3.8 (7.83) | -2.7 (7.64) | -3.8 (11.20) | -2.6 (8.85)
  Delayed memory - Week 52: number analyzed (Participants) | 41 | 22 | 64 | 37
  Delayed memory - Week 52 | -2.0 (8.01) | 3.2 (6.23) | 2.3 (9.09) | 0.6 (11.73)
  CI Delayed memory - Last post baseline assessment: number analyzed (Participants) | 41 | 23 | 0 | 0
  CI Delayed memory - Last post baseline assessment | -1.0 (10.20) | 1.3 (8.44) |  |
  CII Delayed memory - Last on-treatment: number analyzed (Participants) | 0 | 0 | 209 | 141
  CII Delayed memory - Last on-treatment |  |  | -2.5 (10.61) | 0.4 (10.28)
  CII Delayed memory - Last off-treatment: number analyzed (Participants) | 0 | 0 | 169 | 93
  CII Delayed memory - Last off-treatment |  |  | -1.1 (10.75) | 1.1 (11.28)

6. Secondary Outcome: Change in the Everyday Cognition Scale (ECog-Subject) Total Scores
Description: Everyday Cognition Scale (ECog) measures cognitively-relevant everyday abilities comprised of 39 items covering 6 cognitively-relevant domains: Everyday Memory, Everyday Language, Everyday Visuospatial Abilities, Everyday Planning, Everyday Organization, and Everyday Divided Attention. The questionnaire is a self-reported measure completed by both participant and study partner (informant). The total score for the 39 items ranges from 39 to 195, with greater scores indicating worse daily function.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Total scores
Arm/Group | Cohort I (CI) CAD106 | Cohort I (CI) CAD106 Placebo | Cohort II (CII) CNP520 | Cohort II (CII) CNP520 Placebo
Number analyzed (Participants) | 40 | 22 | 178 | 119
Total scores
  Week 26: number analyzed (Participants) | 40 | 22 | 151 | 103
  Week 26 | -1.0 (2.94) | 2.3 (4.80) | 1.8 (6.03) | 0.6 (6.45)
  Week 52: number analyzed (Participants) | 40 | 21 | 63 | 37
  Week 52 | 0.6 (5.23) | 0.4 (2.99) | 2.7 (6.16) | 0.2 (5.01)
  CI Last post baseline assessment: number analyzed (Participants) | 40 | 22 | 0 | 0
  CI Last post baseline assessment | 0.6 (5.02) | 1.6 (4.07) |  |
  CII Last on-treatment: number analyzed (Participants) | 0 | 0 | 178 | 119
  CII Last on-treatment |  |  | 2.6 (7.81) | 0.9 (6.48)
  CII Last off-treatment: number analyzed (Participants) | 0 | 0 | 162 | 86
  CII Last off-treatment |  |  | 1.6 (6.77) | 0.8 (6.13)

7. Secondary Outcome: Change in the Everyday Cognition Scale (ECog-Informant) Total Scores
Description: Everyday Cognition Scale (ECog) measures cognitively-relevant everyday abilities comprised of 39 items covering 6 cognitively-relevant domains: Everyday Memory, Everyday Language, Everyday Visuospatial Abilities, Everyday Planning, Everyday Organization, and Everyday Divided Attention. The questionnaire is a self-reported measure completed by both participant and study partner (informant). The total score for the 39 items ranges from 39 to 195, with greater scores indicating worse daily function. Cohort I=C I and Cohort II=C II.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Total scores
Arm/Group | Cohort I (CI) CAD106 | Cohort I (CI) CAD106 Placebo | Cohort II (CII) CNP520 | Cohort II (CII) CNP520 Placebo
Number analyzed (Participants) | 37 | 23 | 160 | 113
Total scores
  Week 26: number analyzed (Participants) | 37 | 23 | 142 | 95
  Week 26 | -0.4 (4.21) | -1.0 (4.87) | 0.1 (6.84) | -0.7 (8.69)
  Week 52: number analyzed (Participants) | 37 | 22 | 57 | 29
  Week 52 | -0.2 (3.15) | -0.3 (5.12) | 1.4 (5.18) | -0.2 (9.59)
  CI Last post baseline assessment: number analyzed (Participants) | 37 | 23 | 0 | 0
  CI Last post baseline assessment | -1.1 (4.23) | -1.0 (4.88) |  |
  CII Last on-treatment: number analyzed (Participants) | 0 | 0 | 160 | 113
  CII Last on-treatment |  |  | 1.3 (8.76) | 0.1 (9.12)
  CII Last off-treatment: number analyzed (Participants) | 0 | 0 | 143 | 77
  CII Last off-treatment |  |  | 1.4 (8.49) | -0.5 (10.10)

8. Secondary Outcome: Number of Participants With Newly Occurring Safety MRI Abnormalities (ARIA-E, ARIA-H,White Matter Disease and Any Other MRI Abnormalities)
Description: Safety MRI included sequences necessary for ascertainment of possible ARIA-E (Amyloid Related Imaging Abnormality-Edema), ARIA-H (Amyloid Related Imaging Abnormality- Hemorrhage, including superficial siderosis and microhemorrhages), assessment of recent infarcts and white matter integrity examination (White matter disease worsening since baseline) and a general assessment of brain abnormalities. Assessment of cerebral amyloid angiopathy (CAA) is included in the overall safety MRI findings results.
Time Frame: Baseline to end of exposure for a maximum of 1455 days for CI and 907 days for CII
Population: Safety analysis set - only participants with a value at both Baseline and that visit are included. For CI: last post-baseline assessment collected during the study. For CII: Last on-treatment is the last assessment before or at last day on study drug + 31 days. Last off-treatment is the last assessment after last day on study drug + 31 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I (CI) CAD106 | Cohort I (CI) CAD106 Placebo | Cohort II (CII) CNP520 | Cohort II (CII) CNP520 Placebo
Number analyzed (Participants) | 42 | 23 | 249 | 163
Participants
  Questionable presence of ARIA-E | 0 | 0 | 0 | 1
  Presence of ARIA-E | 1 | 0 | 0 | 2
  ARIA-E - If present, the worst Severity=moderate | 1 | 0 | 0 | 2
  Presence of ARIA-H - >4 microhemorrhages (new hemosiderin deposits < 10 mm) | 2 | 0 | 6 | 2
  White matter disease worsening: 1-3 increase | 0 | 2 | 6 | 1
  White matter disease worsening: 4 - 8 increase | 0 | 0 | 0 | 0
  White matter disease worsening > 8 increase | 0 | 0 | 0 | 0
  Any other MRI abnormalities | 2 | 1 | 0 | 0

9. Secondary Outcome: Annualized Percent Change on Volume of Brain Regions
Description: Annualized % change from baseline in volume of specific brain regions of interest (ROIs): whole brain (WB), hippocampus (Hip), and lateral ventricles (LV). Annualized percentage change was calculated as (percentage per participant / time interval (in days)) x 365.25. Time interval (in days) was derived as date of current MRI assessment on study drug - date of baseline MRI assessment + 1.
Time Frame: as for outcome 5
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of volume change
Arm/Group | Cohort I (CI) CAD106 | Cohort I (CI) CAD106 Placebo | Cohort II (CII) CNP520 | Cohort II (CII) CNP520 Placebo
Number analyzed (Participants) | 42 | 23 | 201 | 135
Percentage of volume change
  WB Week 26: number analyzed (Participants) | 35 | 23 | 145 | 104
  WB Week 26 | -0.7570 (1.33114) | -0.6044 (1.29608) | -0.9318 (1.06843) | -0.4616 (1.00537)
  WB Week 52: number analyzed (Participants) | 37 | 22 | 63 | 40
  WB Week 52 | -0.5144 (0.66578) | -0.3395 (0.75810) | -0.6590 (0.64838) | -0.4227 (0.58778)
  WB CI Last post baseline assessment: number analyzed (Participants) | 40 | 23 | 0 | 0
  WB CI Last post baseline assessment | -0.4645 (0.57503) | -0.5321 (0.46526) |  |
  WB CII Last on-treatment: number analyzed (Participants) | 0 | 0 | 148 | 108
  WB CII Last on-treatment |  |  | -0.8268 (0.94889) | -0.5181 (0.92086)
  WB CII Last off-treatment: number analyzed (Participants) | 0 | 0 | 36 | 23
  WB CII Last off-treatment |  |  | -0.6748 (0.62542) | -0.3317 (0.62616)
  Hip Week 26: number analyzed (Participants) | 35 | 23 | 145 | 104
  Hip Week 26 | -1.3262 (2.35453) | -0.9245 (2.81731) | -1.6603 (2.65529) | -0.8817 (2.06227)
  Hip Week 52: number analyzed (Participants) | 37 | 22 | 63 | 40
  Hip Week 52 | -1.0376 (1.44310) | -0.7780 (1.81604) | -1.2438 (1.79988) | -0.9567 (1.42941)
  Hip CI Last post baseline assessment: number analyzed (Participants) | 40 | 23 | 0 | 0
  Hip CI Last post baseline assessment | -1.0801 (1.38061) | -1.0477 (1.33603) |  |
  Hip CII Last on-treatment: number analyzed (Participants) | 0 | 0 | 148 | 108
  Hip CII Last on-treatment |  |  | -1.4790 (2.36526) | -0.9984 (1.85655)
  Hip CII Last off-treatment: number analyzed (Participants) | 0 | 0 | 36 | 23
  Hip CII Last off-treatment |  |  | -1.9375 (2.03593) | -1.0498 (1.66596)
  LV Week 26: number analyzed (Participants) | 35 | 23 | 145 | 104
  LV Week 26 | 4.1848 (5.77286) | 2.5581 (7.54667) | 4.5176 (5.59748) | 3.9735 (4.23237)
  LV Week 52: number analyzed (Participants) | 37 | 22 | 63 | 40
  LV Week 52 | 4.2060 (3.92877) | 2.8232 (5.04358) | 3.3854 (3.71214) | 2.9059 (3.18734)
  LV CI Last post baseline assessment: number analyzed (Participants) | 40 | 23 | 0 | 0
  LV CI Last post baseline assessment | 4.0543 (3.75310) | 3.5427 (3.53772) |  |
  LV CII Last on-treatment: number analyzed (Participants) | 0 | 0 | 148 | 108
  LV CII Last on-treatment |  |  | 4.3588 (5.07839) | 4.0308 (3.64102)
  LV CII Last off-treatment: number analyzed (Participants) | 0 | 0 | 36 | 23
  LV CII Last off-treatment |  |  | 3.9617 (2.61831) | 2.6052 (3.54903)

10. Secondary Outcome: Change in Cerebrospinal Fluid (CSF) Levels of Amyloid Beta 40 (Aβ40)
Description: Alzheimer's Disease-related biomarkers analyzed in cerebrospinal fluid (CSF): Amyloid Beta 40 (Aβ40)
Time Frame: Baseline to last assessment
Population: No lumbar punctures for CSF collection were performed due to early termination of trial
Arm/Group | Cohort I (CI) CAD106 | Cohort I (CI) CAD106 Placebo | Cohort II (CII) CNP520 | Cohort II (CII) CNP520 Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Change in Cerebrospinal Fluid (CSF) Levels of Amyloid Beta 42 (Aβ42)
Description: Alzheimer's Disease-related biomarkers analyzed in cerebrospinal fluid (CSF): Amyloid Beta 42 (Aβ42)
Time Frame: Baseline to last assessment
Population: No lumbar punctures for CSF collection were performed due to early termination of trial
Arm/Group | Cohort I (CI) CAD106 | Cohort I (CI) CAD106 Placebo | Cohort II (CII) CNP520 | Cohort II (CII) CNP520 Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Change in Cerebrospinal Fluid (CSF) Levels of Total Tau and Phosphorylated Tau
Description: Alzheimer's Disease-related biomarkers analyzed in cerebrospinal fluid (CSF): total tau protein and phosphorylated tau protein levels
Time Frame: Baseline to last assessment
Population: No lumbar punctures for CSF collection were performed due to early termination of trial
Arm/Group | Cohort I (CI) CAD106 | Cohort I (CI) CAD106 Placebo | Cohort II (CII) CNP520 | Cohort II (CII) CNP520 Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Change in Neurofibrillary Tangle Burden as Measured by Standardized Uptake Ratio (SUVR) of PET Scans With Tau Radiotracer (Where Available)
Description: To demonstrate the effects of CNP520 vs placebo on tau pathology in the brain
Time Frame: Baseline to last assessment
Population: No post baseline data collected
Arm/Group | Cohort I (CI) CAD106 | Cohort I (CI) CAD106 Placebo | Cohort II (CII) CNP520 | Cohort II (CII) CNP520 Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Cohort I : Annualized Change in Amyloid Deposition as Measured by Centiloids of Positron Emission Tomography (PET) Scan With Amyloid Radiotracer
Description: To demonstrate the effects of CAD106 vs placebo on Alzheimer's Disease-related biomarkers
Time Frame: Baseline up to approximately Week 104
Population: Only available for Cohort I. For Cohort II, no post-baseline (year 2) amyloid PET scans could be obtained due to the early trial termination
Measure: Mean (Standard Deviation); unit: Centiloids
Arm/Group | Cohort I (CI) CAD106 | Cohort I (CI) CAD106 Placebo
Number analyzed (Participants) | 42 | 23
Centiloids | -0.911 (5.6596) | 8.367 (6.6805)

15. Secondary Outcome: Change in Serum Neurofilaments
Description: Alzheimer's Disease-related biomarkers analyzed in blood serum: light chain neurofilaments (NfL)
Time Frame: Baseline to Week 26 and week 52, CI baseline to last assessment. CII baseline to last on-treatment and to last off-treatment
Population: Only participants with a value at both Baseline and that visit are included. CI last post-baseline assessment. CII Last on-treatment is the last assessment before or at last day on study drug + 31 days.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cohort I (CI) CAD106 | Cohort I (CI) CAD106 Placebo | Cohort II (CII) CNP520 | Cohort II (CII) CNP520 Placebo
Number analyzed (Participants) | 20 | 10 | 72 | 53
pg/mL
  Week 26 | 1.44 (3.165) | -3.89 (13.058) | 0.644 (3.4879) | 0.362 (6.7547)
  Week 52: number analyzed (Participants) | 8 | 6 | 8 | 9
  Week 52 | 2.63 (5.716) | -6.09 (16.542) | 1.921 (4.0515) | -4.852 (14.2270)
  C I Last post baseline assessment: number analyzed (Participants) | 20 | 10 | 0 | 0
  C I Last post baseline assessment | 1.77 (4.643) | -3.31 (12.858) |  |
  C II Last on-treatment: number analyzed (Participants) | 0 | 0 | 72 | 51
  C II Last on-treatment |  |  | 0.647 (3.5357) | 0.280 (6.8289)
  C II Last off-treatment: number analyzed (Participants) | 0 | 0 | 2 | 2
  C II Last off-treatment |  |  | -0.004 (3.7102) | -2.145 (2.6799)

16. Secondary Outcome: Number of Suicidal Ideation or Behavior Events
Description: Prospective suicidality assessment was performed with the use of Columbia-Suicide Severity Rating Scale (C-SSRS), a questionnaire using a detailed branched logic algorithm evaluating participant's suicidality ideation and behavior. Answer "yes" on item 4 or 5 of the Suicidal Ideation section or "yes" on any item of the Suicidal Behavior section was considered positive.
Time Frame: Baseline to end of exposure for a maximum of 1455 days for CI and 907 days for CII
Population: Safety analysis set which includes only participants with events
Measure: Number; unit: events
Arm/Group | Cohort I (CI) CAD106 | Cohort I (CI) CAD106 Placebo | Cohort II (CII) CNP520 | Cohort II (CII) CNP520 Placebo
Number analyzed (Participants) | 42 | 23 | 249 | 163
events
  Any suicidal ideation | 2 | 1 | 12 | 4
  Any suicidal behavior | 0 | 0 | 1 | 1

17. Secondary Outcome: Cohort I : Change in Cognition as Measured by APCC and CDR-SOB Scores and Antibody Response
Time Frame: Month 6 to Month 60
Population: No analysis performed due to early termination, no month 60 data
Arm/Group | Cohort I (CI) CAD106 | Cohort I (CI) CAD106 Placebo | Cohort II (CII) CNP520 | Cohort II (CII) CNP520 Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

18. Secondary Outcome: Cohort I: Peak Concentration (Cmax) of CAD106 Induced Abeta-specific Antibody Titers
Description: Cmax is the maximum Titer Concentration of any post-baseline 'on treatment' visit. A visit is considered as 'on treatment' if visit date is within {last injection + 180 days}.
  - Geometric mean and CI's are back-transformed from the estimates for Log mean and CI's.
Time Frame: Week 9, 13, 15, 26 and quarterly thereafter (trough values)
Population: Safety population
Measure: Geometric Mean (95% Confidence Interval); unit: Days x titer levels rel. to ref. serum
Arm/Group | Cohort I (CI) CAD106
Number analyzed (Participants) | 41
Days x titer levels rel. to ref. serum | 128.76 [99.05 to 167.37]

19. Secondary Outcome: Cohort I: Area Under the Concentration Curve (AUC) of CAD106 Induced Abeta-specific Antibody Titers
Description: AUC is calculated based on 'on treatment' visit only.(missing values for peak visits were linearly interpolated for calculation; missing values for trough visits were imputed by average of non-missing trough values.).
Time Frame: Week 9, 13, 15, 26 and quarterly thereafter (trough values)
Population: Safety population
Measure: Geometric Mean (95% Confidence Interval); unit: Days x titer levels rel. to ref. serum
Arm/Group | Cohort I (CI) CAD106
Number analyzed (Participants) | 42
Days x titer levels rel. to ref. serum | 34999.89 [22992.17 to 53278.68]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment plus 31 days of washout period for a maximum duration of 1455 days for CI and 907 days for CII
Groups:
- Cohort I @CAD106: Cohort I @CAD106
- Cohort I @Placebo: Cohort I @Placebo
- Cohort II (CNP520 50): CNP520 (50 mg) capsules taken once daily orally
- Cohort II Placebo: Cohort II @Placebo
Arm/Group | Cohort I @CAD106 | Cohort I @Placebo | Cohort II (CNP520 50) | Cohort II Placebo
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/23 | 0/249 | 0/163
Serious Adverse Events (participants affected / at risk) | 4/42 | 3/23 | 8/249 | 7/163
Other Adverse Events (participants affected / at risk) | 36/42 | 21/23 | 106/249 | 76/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort I @CAD106 (N=42) | Cohort I @Placebo (N=23) | Cohort II (CNP520 50) (N=249) | Cohort II Placebo (N=163)
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Feeling jittery (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebellar haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort I @CAD106 (N=42) | Cohort I @Placebo (N=23) | Cohort II (CNP520 50) (N=249) | Cohort II Placebo (N=163)
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 1
Type V hyperlipidaemia (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Deafness bilateral (Ear and labyrinth disorders) | 2 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 0 | 3 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0 | 0 | 0
Thyroid mass (Endocrine disorders) | 0 | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 0 | 7 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 6 | 3
Eosinophilic oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 5 | 4
Pancreatic cyst (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Salivary gland disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 2 | 0 | 0 | 0
Fatigue (General disorders) | 11 | 1 | 3 | 1
Influenza like illness (General disorders) | 5 | 0 | 0 | 0
Injection site erythema (General disorders) | 1 | 1 | 0 | 0
Injection site pain (General disorders) | 10 | 0 | 0 | 0
Injection site pruritus (General disorders) | 2 | 0 | 0 | 0
Injection site reaction (General disorders) | 4 | 0 | 0 | 0
Malaise (General disorders) | 3 | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 7 | 1 | 4 | 0
Seasonal allergy (Immune system disorders) | 2 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 2 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 1 | 1 | 8
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1
Conjunctivitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Dacryocanaliculitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 1 | 1
Influenza (Infections and infestations) | 1 | 2 | 3 | 0
Nasopharyngitis (Infections and infestations) | 4 | 2 | 10 | 2
Pharyngitis (Infections and infestations) | 1 | 1 | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 3 | 1 | 5 | 8
Upper respiratory tract infection (Infections and infestations) | 7 | 3 | 11 | 11
Urinary tract infection (Infections and infestations) | 0 | 2 | 5 | 4
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 4
Contusion (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 3
Fall (Injury, poisoning and procedural complications) | 4 | 1 | 8 | 4
Injection related reaction (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Mallet finger (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0
Lumbar puncture (Investigations) | 0 | 1 | 0 | 0
Urine albumin/creatinine ratio increased (Investigations) | 0 | 0 | 9 | 2
Weight decreased (Investigations) | 0 | 0 | 7 | 1
Weight increased (Investigations) | 2 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 2 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 6 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 7 | 6
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 5 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 3 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2 | 6 | 5
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 2
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 1 | 0 | 0
Cerebral cyst (Nervous system disorders) | 0 | 1 | 0 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 7 | 1
Headache (Nervous system disorders) | 7 | 0 | 6 | 9
Lethargy (Nervous system disorders) | 2 | 0 | 2 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 2 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 2 | 1 | 19 | 5
Anxiety (Psychiatric disorders) | 0 | 0 | 11 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 4 | 9
Irritability (Psychiatric disorders) | 1 | 1 | 2 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 1 | 0 | 0
Hypercalciuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 5 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 10 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Essential hypertension (Vascular disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated due to unexpected changes in cognitive function, brain volume loss, and body weight loss. Cohort II (CNP520) treatment was stopped and evaluated through an off-treatment follow-up period. After the decision to terminate Cohort II of the study (CNP520), treatment with CAD106 (Cohort I) was also terminated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/11/NCT02565511/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/11/NCT02565511/SAP_001.pdf